CLINICAL TRIAL: NCT05157984
Title: Evaluation of Peroral Endoscopic Myotomy to Treat Zenker's Diverticulum
Acronym: ZPOEM
Status: Enrolling by invitation | Type: Observational
Sponsor: Methodist Health System (Other)
Collaborators: Baylor Scott and White Health (Other)
Responsible Party: Sponsor
Other Study IDs: 031.GID.2021.D; 2020.11.16 (Other: Baylor Scott and White)
Record Dates: First submitted 2021-06-10; First posted 2021-12-15 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Zenker Diverticulum
Keywords: Zenker's Diverticulum; peroral endoscopic myotomy
MeSH Terms: conditions — Zenker Diverticulum

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Retrospective cohort: Any patient of the physicians listed in this study who has undergone the ZPOEM procedure to treat ZD at Methodist Health System
  Interventions: Procedure: ZPOEM
- Prospective cohort: Any patient of the physicians listed in this study who has undergone the ZPOEM procedure to treat ZD at Methodist Health System and has agreed to be follow-up post-procedure.
  Interventions: Procedure: ZPOEM

INTERVENTIONS:
Procedure: ZPOEM — Zenker's diverticulum management by Per oral endoscopic myotomy (POEM)
  Other Names: peroral endoscopic myotomy (POEM)

SUMMARY:
This is a multicenter investigator-initiated trial between Baylor-Scotts & White (BSW) and Methodist Health System (MHS). This study will be conducted via a retrospective review and a prospective patient registry. Patients who have undergone the ZPOEM procedure performed by the physicians listed in this protocol will be included, as well as patients who will have this procedure in the future. Data that will be collected at MHS will be entered into an Excel spreadsheet. Patient demographic information will be collected via a review of subjects' electronic medical records. Available patient outcomes will be collected via a review of electronic medical records. This review will be conducted from 1/1/2017 through 12/31/2025.

DETAILED DESCRIPTION:
This is a multicenter investigator-initiated trial between Baylor-Scotts & White (BSW) and Methodist Health System (MHS). This study will be conducted via a retrospective review and a prospective patient registry. Patients who have undergone the ZPOEM procedure performed by the physicians listed in this protocol will be included, as well as patients who will have this procedure in the future. Data that will be collected at MHS will be entered into an Excel spreadsheet. Patient demographic information will be collected via a review of subjects' electronic medical records. Available patient outcomes will be collected via a review of electronic medical records. This review will be conducted from 1/1/2017 through 12/31/2025.

To obtain the follow-up information, potential subjects will be identified using the same process described in the previous paragraph and will be contacted by a member of the institution's research team to answer questions about their symptoms post-surgery. These are listed in the ZPOEM Data Collection Sheet. These questions may be administered over the phone, via email, or by mail. Subjects enrolled in the patient registry will have follow-up data collected at 2-time points: 2 weeks post-op and 3 months post-op.

Primary endpoints and other variables to be collected are those listed on the ZPOEM Data Collection Sheet. Primary subject endpoints include, but are not limited to:

* Dysphagia score(s) - depending on what is available in EMR
* Weight gain following surgery

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age or older
* Any patient of the physicians listed in this study who has undergone the ZPOEM procedure to treat ZD at MHS
* For prospective registry: Ability to give informed consent

Exclusion Criteria:

* For prospective registry: Unable or not willing to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with Zenker's diverticulum (ZD) and who have undergone the ZPOEM procedure, as well as patients who will have this procedure in the future
Sampling Method: Non-Probability Sample
Enrollment: 38 (Estimated)
Dates: Start 2021-06-25 (Actual); Primary Completion 2024-06-28 (Estimated); Study Completion 2024-06-28 (Estimated)

PRIMARY OUTCOMES:
Retrospective chart review / Compartive analyses; t-tests and Wilcoxon-Mann-Whiteney Test; Chi-square or Fisher's exact test; and Pearson correlation coeffecient or Spearman's rank-order correlation | January 2017 to December 2025
  Retrospective review of patient records who have had ZPOEM procedure, compartive analyses will be performed by employing statistical tests such as t-tests and Wilcoxon-Mann-Whiteney Test; Chi-square or Fisher's exact test; and Pearson correlation coeffecient or Spearman's rank-order correlation depdening on the data distribution. Multivariate analyses will be employed with a p-value <0.05 will indicate statistical significance.

SECONDARY OUTCOMES:
Prospective follow-up of patients/ Compartive analyses; t-tests and Wilcoxon-Mann-Whiteney Test; Chi-square or Fisher's exact test; and Pearson correlation coeffecient or Spearman's rank-order correlation | June 2021 to December 2025
  Follow up of patients who had the ZPOEM procedure / Compartive analyses will be performed by employing statistical tests such as t-tests and Wilcoxon-Mann-Whiteney Test; Chi-square or Fisher's exact test; and Pearson correlation coeffecient or Spearman's rank-order correlation depdening on the data distribution. Multivariate analyses will be employed with a p-value <0.05 will indicate statistical significance.

CONTACTS AND LOCATIONS:
Overall Officials: Prashant Kedia, MD, Principal Investigator — Methodist Health System
Locations (1):
- Methodist Dallas Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No
Participant data will be shared only with Baylor, Scott & White. All data will be de-identified and in compliance with the Data User Agreement in place between both institutions.